CLINICAL TRIAL: NCT04711317
Title: Pre-oxygenation With High-flow Nasal Cannula in Pregnant Women Undergoing Caesarian Section Under General Anesthesia - a Pilot Study
Brief Title: Pre-oxygenation With High-flow Nasal Cannula in Caesarian Section Under General Anesthesia
Acronym: PRIOROB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Danderyds Hospital, Stockholm, Sweden (Unknown); Stockholm South General Hospital (Other); Karlstad Central Hospital (Other); Östra Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, Senior Consultant, Associate Professor, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIOROB
Record Dates: First submitted 2020-12-09; First posted 2021-01-15 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related; Anesthesia; Oxygen Deficiency; Cesarean Section Complications
Keywords: Preoxygenation; Perioxygenation; Nasal high flow oxygen; Cesarian sectio
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: One intervention group that is compared to a control group that is standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoxygenation with nasal high flow oxygen (Experimental): Preoxygenation with nasal high flow oxygen
  Interventions: Device: Nasal high flow oxygen
- Control group (No Intervention): Standard preoxygenation according to hospital protocol with tight fitting facemask

INTERVENTIONS:
Device: Nasal high flow oxygen — Pregnant women scheduled for cesarian section in general anaesthesia will be preoxygenated using nasal high flow oxygen
  Arms: Preoxygenation with nasal high flow oxygen

SUMMARY:
The investigators and other groups have demonstrated that high-flow nasal oxygen used during preoxygenation for emergency surgery is at least equally effective as preoxygenation compared to standard tight fitting mask. The investigators also have data from a recent study that indicates that high-flow nasal oxygen might decrease the risk of clinically relevant desaturation below 93% of arterial oxygen saturation.

The studies investigating the concept of high-flow nasal oxygen has up to this date excluded pregnant women. Pregnant woman is a patient group with known difficulties to maintain adequate saturation levels during apnoea. Due to smaller functional residual capacity their oxygen stores after preoxygenation are smaller compared to patients with a normal body mass index. The pregnant woman also have a higher oxygen demand and metabolism due to the growing placenta and the fetus. Pregnant women are therefore a patient group where a method that could prolong time until desaturation would be even more valuable and potentially could save lives.

Based on the above, the investigators now aim to conduct a clinical pilot study, where pregnant women undergoing caesarian section under general anesthesia are pre and perioxygenated with high-flow nasal oxygen. Data from that group will be compared with patients preoxygenated in a traditional manner with tight facemask. This study is done to evaluate an established technique on a patient category that in theory could gain a lot from it.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, >18 years old
2. Caesarian section under general anesthesia.
3. Pregnant in week 30 or later
4. Capable of understanding the study information and signing the written consent.

Exclusion Criteria:

1. BMI >45
2. Dependency on non-invasive ventilation to maintain oxygen saturation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with peripheral arterial oxygen saturation below 93% from start of pre-oxygenation until one minute after tracheal intubation and comparison between intervention and control | Up to 1 minute after intubation
  arterial peripheral oxygen saturation

SECONDARY OUTCOMES:
Comparison of Endtidal concentration of oxygen after intubation between intervention and control | The first breaths after intubation eg. within 20 seconds of intubation
Comparison of Endtidal carbondioxide concentration after intubation between intervention and control | The first breaths after intubation eg. within 20 seconds of intubation
Comparison of Number of patients with regurgitation of gastric contents between intervention and control | During intubation eg up to 0 seconds after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital and Karolinska Insitutet
Locations (4):
- Sweden (4):
  - Karlstads Centralsjukhus, Karlstad
  - Danderyds Hospital, Stockholm
  - Karolinska University Hospital, Solna, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No